CLINICAL TRIAL: NCT00302354
Title: A Double-blind Randomized, Placebo-controlled, Crossover Study of Single Doses of OROS Methylphenidate Hydrochloride (CONCERTA) and Long-acting Methylphenidate Hydrochloride (RITALIN LA) in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Thomas J. Spencer, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2004-P-002212
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Volunteers

INTERVENTIONS:
Drug: OROS methylphenidate HCl
Drug: SODAS methylphenidate HCl

SUMMARY:
This is a double-blind, placebo-controlled study, three-period crossover study to examine the likeability of a single dose of OROS MPH (CONCERTAÒ 90mg) and a single dose of Long-acting MPH (RITALIN LAÒ 90mg). Hypotheses are as follows:

Hypothesis 1: OROS-MPH (CONCERTAÒ) will be later than SODOS-MPH (RITALIN LAÒ) in its Tmax (time to Cmax).

Hypothesis 2: The subjective feelings of detection and likeability would be greater for SODOS-MPH (RITALIN LAÒ) than for an equivalent total dose of OROS-MPH (CONCERTAÒ).

DETAILED DESCRIPTION:
Our recent work has suggested that the potential euphoriant risk associated with MPH may be moderated by the oral delivery system in which a longer delivery system may be safer than the immediate release one. OROS-MPH's pharmacokinetic profile uses an increasing delivery of MPH over the day (ascending pharmacokinetic curve). It was designed to replace IR-MPH TID treatment. Another new long-acting MPH formulation is the spheroidal oral drug absorption system (SODAS). SODAS-MPH consists of capsules with two types of beads in a 1 to 1 ratio. Evaluating whether different long acting formulations of MPH will differ in their rate of onset of MPH action (plasma level) is of high clinical, scientific and public health relevance. Since the rate of delivery of MPH is a key factor previously associated with detection and likeability of MPH.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females. With the exception of women who have been post-menopausal for a minimum of 12 months prior to screening and those who have undergone hysterectomy or bilateral oophorectomy, all female subjects must have a negative urine pregnancy test at both screening and at each admission to the research unit, and have used a medically acceptable form of birth control for at least one month prior to screening and willing to continue use during the study. Medically acceptable forms of birth control include abstinence, hormonal contraceptives, diaphragm with spermicide, condom with spermicide, intrauterine device, or surgical sterilization (including vasectomy of male partner(s).
2. Eighteen (18) to 45 years of age, inclusive.
3. Based on medical history, physical examination, and/or lab results, are considered healthy and free of any conditions that may interfere with participation in the study. Any abnormalities at screening on results of ECG or any laboratory test must be determined to be not clinically significant by the investigator.
4. Agree to not use prescription stimulants (except for the study medication) during the study.
5. Have venous access sufficient for blood sampling as determined by clinical examination.
6. Weigh at least 110 pounds at screening.
7. Agree and are available to return to the study center for three full-day (approximately 14 hours) study visits held five to 30 days apart within a 10-week period, and willing to complete all protocol-specified assessments.
8. Able to read and comprehend English

Exclusion Criteria:

1. Known hypersensitivity to methylphenidate or components of CONCERTA or RITALIN, or to the sympathomimetic amines.
2. Presence or history of any medically diagnosed, clinically significant Axis I psychiatric disorder (including substance use disorders, bipolar disorder, any psychotic disorder, Tourette's disorder or family history of Tourette's)
3. Any clinically significant chronic disease or unstable medical abnormality by history or physical examination, including hypertension, glaucoma, hyperthyroidism, a seizure disorder, history of myocardial infarction or stroke, or history of cardiac arrhythmia or heart murmur (other than uncomplicated mitral valve prolapse).
4. Clinically significant abnormal baseline laboratory values which include the following:

   1. Values > 20% above the upper range of the laboratory standard of a basic metabolic screen.
   2. Exclusionary blood pressure > 140 (systolic) and 95 (diastolic).
   3. Exclusionary ECG parameters: QTC > 460 msec, QRS > 120 msec, and PR > 200 msec. Subjects having ECG evidence of ischemia or arrhythmia as reviewed by an independent cardiologist.
5. Currently taking a monoamine oxidase inhibitor or have taken a monoamine oxidase inhibitor in the 14 days before initiation of study medication.
6. Currently taking or require any of the following medications: clonidine or other alpha-2 adrenergic receptor agonists, tricyclic antidepressants, selective serotonin reuptake inhibitors (SSRIs), theophylline, coumarin anticoagulants, anticonvulsants, or prescription stimulants.
7. Have taken an SSRI in the 35 days before initiation of the study medication.
8. Currently physically dependent on benzodiazepines, opiates or alcohol as determined by clinical evaluation or positive urine drug screen at screening.
9. Preexisting severe gastrointestinal narrowing (pathologic or iatrogenic, for example: small bowel inflammatory disease, "short gut" syndrome due to adhesions or decreased transit time, past history of peritonitis, cystic fibrosis, chronic intestinal pseudoabsorption, or Meckel's diverticulum).
10. Unable to swallow the study medication whole.
11. Have had a significant blood loss (>500 mL) or donated blood in the 30 days preceding dosing.
12. Have a positive urine drug screen at screening.
13. Have taken an investigational medication or product within the past 30 days.
14. Have taken prescription medications (with the exception of birth control methods) within seven days of screening or is anticipated to need any medications, over-the- counter products (other than acetaminophen), or herbal supplements during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2004-12; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Objective measures provided by hourly d and l ritalinic acid and methylphenidate levels from pre-dose and hours 1,2,3,4,5,6,7,8,10, and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States